CLINICAL TRIAL: NCT06274502
Title: Automated Detection and Diagnosis of Pathological DRGs in PHN Patients Using Deep Learning and Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: deep learning
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Deep Learning
Keywords: deep learning; Magnetic resonance neurography; dorsal root ganglion; postherpetic neuralgia; YOLOv8
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: YOLOv8 — After image post-processing, the You Only Look Once (YOLO) version 8 was selected as the target algorithm model.

SUMMARY:
Here, this study aimed to develop an automated system for detecting and diagnosing lesion DRGs in PHN patients based on deep learning. This study retrospectively analyzed the DRG images of all patients with postherpetic neuralgia who underwent magnetic resonance neuroimaging examinations in our radiology department from January 2021 to February 2022. After image post-processing, the You Only Look Once (YOLO) version 8 was selected as the target algorithm model. Model performance was evaluated using metrics such as precision, recall, Average Precision, mean average precision and F1 score.

DETAILED DESCRIPTION:
Our previous research has confirmed differences in macroscopic and microscopic aspects between the imaging of lesioned dorsal root ganglia (DRG) in patients with postherpetic neuralgia (PHN) and healthy controls. Additionally, our study revealed that while lesioned skin localization is a classic method in clinical practice, there is still a certain rate of discrepancy with the lesioned DRG observed in magnetic resonance imaging (MRI). This suggests the significant value of MRI in diagnosing lesioned DRG in PHN patients. For patients with zoster sine herpete neuralgia, it is even more crucial to identify the lesioned DRG through MRI. However, due to the small size and varied morphology of DRG lesions, diagnosing lesioned DRG through MRI requires specialized knowledge in neuroanatomy and imaging, posing a challenge to clinical practitioners. Identifying lesioned DRG rapidly and accurately is crucial for interventional therapy, as it serves as an essential treatment target for neuropathic pain.

The YOLO (You Only Look Once) series of algorithms are currently widely used single-stage real-time object detection algorithms, including YOLOv1-YOLOv8. Due to their extremely high detection speed, they enable real-time object detection. YOLOv5 and YOLOv8 are now extensively employed in various applications such as autonomous driving, video surveillance, and object tracking. Moreover, the YOLO series is increasingly being applied in the medical field, including tumor and joint capsule lesion detection, demonstrating good accuracy, recall rates, and detection efficiency. This study aims to utilize the YOLOv8 algorithm to develop a fast and accurate object detection model, simultaneously evaluating its performance. It seeks to validate the feasibility and effectiveness of detecting lesioned dorsal root ganglia (DRG) in real-time postherpetic neuralgia using this model, providing a basis for early diagnosis for clinical practitioners and enabling rapid and precise localization of lesioned DRG.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Patients with herpes zoster who continue to experience pain for over one month after the crust forms over the skin lesions;
* Clear MRI images showing evident dorsal root ganglia (DRG) lesions.

Exclusion Criteria:

* Patients with severe systemic, metabolic, or neurological diseases that can lead to polyneuropathy, such as multiple myeloma, diabetes, or thyroid diseases;
* Patients with a history of psychiatric disorders, other chronic pain conditions, or substance abuse;
* Patients with a history of thoracic or back surgeries and a history of pain;
* Presence of artifacts in the imaging or unclear image display;
* Target images obscured by other tissues.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postherpetic neuralgia due who underwent magnetic resonance neuroimaging examinations in the Radiology Department at our hospital from January 2021 to February 2022.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Develop an automated system for detecting and diagnosing lesion DRGs in PHN patients based on deep learning | 202310-202402
  the You Only Look Once (YOLO) version 8 was selected as the target algorithm model

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided